CLINICAL TRIAL: NCT00637572
Title: A Randomized, Open-labeled, Pilot Study Comparing Weight Gain in Adults With AIDS-related Wasting Given Either Megestrol Acetate Oral Suspension Nanocrystal Dispersion (MA-NCD) or Megestrol Acetate Oral Suspension (Megace)
Brief Title: Evaluate Weight Gain Using 2 Different Formulations of Megestrol Acetate Oral Suspension for AIDS-related Weight Loss
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAR-002
Record Dates: First submitted 2008-03-11; First posted 2008-03-18 (Estimated); Results first posted 2016-04-20 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-09

CONDITIONS: HIV Infections; Cachexia; Anorexia; AIDS Wasting Syndrome; HIV Wasting Syndrome
Keywords: Weight loss; Cachexia; Anorexia; Megestrol acetate oral suspension; Nanocrystal dispersion; Nanocrystal technology; Body weight changes; AIDS wasting; HIV wasting; Emaciation; Megace ES; Megace; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Cachexia; Anorexia; HIV Wasting Syndrome; Weight Loss; Body Weight Changes; Emaciation | interventions — Megestrol Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Megestrol acetate oral suspension nanocrystal dispersion (Experimental): Megestrol acetate oral suspension nanocrystal dispersion formulation 115 mg/mL
  Interventions: Drug: Megestrol acetate oral suspension nanocrystal dispersion 115 mg/mL
- Megestrol acetate oral suspension micronized formulation (Active Comparator): Megestrol acetate oral suspension micronized formulation 60 mg/mL
  Interventions: Drug: Megestrol acetate oral suspension 40 mg/mL

INTERVENTIONS:
Drug: Megestrol acetate oral suspension nanocrystal dispersion 115 mg/mL — Megestrol acetate oral suspension nanocrystal dispersion 115 mg/mL administered as 575 mg once per day (5 mL dose)
  Other Names: Megace ES
  Arms: Megestrol acetate oral suspension nanocrystal dispersion
Drug: Megestrol acetate oral suspension 40 mg/mL — Megestrol acetate oral suspension 40 mg/mL administered as 800 mg once per day (20 mL dose)
  Other Names: Megace
  Arms: Megestrol acetate oral suspension micronized formulation

SUMMARY:
Explore weight gain in HIV-positive patients who have weight loss associated with AIDS-related wasting (anorexia/cachexia). Patients are treated for 12 weeks with either megestrol acetate oral suspension nanocrystal dispersion formulation, or megestrol acetate oral suspension original formulation

ELIGIBILITY:
Inclusion Criteria:

* Capable of and willing to provide informed consent
* Evidence of HIV infection (either HIV-seropositive, CD4+ T-cell count of ≤350/mm3 or other clinically accepted indicator)
* An unintentional weight loss resulting in a weight 10% less than the lower limit of Ideal Body Weight for frame size, or a recent history of unintentional weight loss of 10% from the subjects baseline
* Weight losses was clinically associated with AIDS-related wasting and not related to any other disease process
* Women of childbearing potential had to agree to use effective contraception for the duration of the study and for two weeks after the last dose
* Clinical laboratory values had to be within normal limits or out-of-range limits must be designated as not clinically significant (some exceptions per protocol)
* Able to read and write in the study related documents translated into the primary local language
* Capable of and willing to return to the clinic regularly for study visits
* Must have been taking a stable regimen of accepted HIV anti-retroviral treatments for at least two weeks prior to study entry
* Capable of completing a 3-day food intake diary with instruction
* Willing to abstain from any illegal or recreational drug substances for the duration of the trial
* Willing to abstain from taking any other medications or substances known to affect appetite or weight gain (eg, steroids [other than those inhaled for treatment of asthmatic conditions], nutritional supplements [other than vitamins or minerals], dronabinol, recombinant human growth hormone, etc.)

Exclusion Criteria:

* Weight loss due to factors other than AIDS-related wasting
* Enrollment in any other clinical trial
* Lack of access to regular meals
* Women of childbearing potential could not be pregnant or nursing
* Clinically severe depression evidenced by a baseline score of 17 or more on the Hamilton Depression Rating Scale (GRID-HAMD-17)
* Recent evidence of or history of significant psychiatric illness that may have compromised the subject's ability to comply with the study requirements
* Intractable or frequent vomiting that regularly interfered with eating
* Clinically significant diarrhea that would have interfered with absorption of foods or medications
* Clinically significant oral lesions or dental conditions that would have interfered with eating a regular diet
* History or evidence of thromboembolic events or any first degree relative with a history of thromboembolic events
* Active AIDS-defining illness or other clinically significant or uncontrolled medical problems
* Current evidence of or history of diabetes mellitus or hypoadrenalism
* Systemic treatment with glucocorticoids within the 12 months prior to study entry

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2004-12; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Fourie, MD, Principal Investigator — 58 Ann Street, Dundee, KZ-Natal 3000, S. Africa
Locations (12):
- Drexel University College of Medicine, Philadelphia, Pennsylvania, United States
- India (4):
  - Victoria Hospital, Bangalore, Karnataka
  - M.S. Ramaiah Medical College and Hospital, Bangalore, Karnataka
  - Kasturba Medical College, Mangalore, Karnataka
  - Ruby Hall Clinic and Grant Medical Foundation, Pune, Maharashtra
- South Africa (7):
  - St Mary's Hospital, Private Bag, Ashwood
  - Quinta-research, Pellissier, Bloemfontein
  - Genclin Corporation, Clinical Trial Centre, Westdene, Bloemfontein
  - 40 Arthur Hobbs Street, Boksburg, Johannesburg
  - 6 Calypso Centre, Richards Bay, KwaZulu-Natal
  - Eastmed Hospital, Eastlynn, Pretoria
  - TrialTech Clinical Research, Hatfield, Pretoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wanke C; Gutierrez J; Kristensen A; MacEarchern L. Safety and efficacy of two preparations of megestrol acetate in HIV-infected individuals with weight loss in Africa, India, and the United States. J Applied Res 2007;7(3):206-216
- See also: Link to published study — http://jrnlappliedresearch.com/articles/index.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Megestrol Acetate Oral Suspension Nanocrystal Dispersion: Subjects were treated with 575 mg per day as single-dose for 12 weeks
- Megestrol Acetate Oral Suspension Micronized Formulation: Subjects were treated with 800 mg per day as single-dose for 12 weeks
Period: Overall Study
Arm/Group | Megestrol Acetate Oral Suspension Nanocrystal Dispersion | Megestrol Acetate Oral Suspension Micronized Formulation
Started | 32 | 31
Completed | 29 | 24
Not Completed | 3 | 7
Not completed — Adverse Event | 1 | 2
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Illicit Drug Use | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis based on Intend to Treat (ITT) population; all randomized subjects who were dispensed medication and had at least one post-randomization visit.
Groups:
- Megestrol Acetate Oral Suspension Nanocrystal Dispersion: Subjects were treated with 575 mg per as single-dose for 12 weeks
- Megestrol Acetate Oral Suspension Micronized Formulation: Subjects were treated with 800 mg per as single-dose for 12 weeks
- Total: Total of all reporting groups
Arm/Group | Megestrol Acetate Oral Suspension Nanocrystal Dispersion | Megestrol Acetate Oral Suspension Micronized Formulation | Total
Number analyzed (Participants) | 32 | 31 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (7.32) | 36.3 (7.22) | 36.8 (7.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 16 | 27
  Male | 21 | 15 | 36

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight
Description: Weight gain in adult HIV positive subjects who have weight loss with AIDS related wasting within the first 12 weeks of treatment
Time Frame: Baseline (Day 1) to Week 12
Population: Analysis is based on Intent-To-Treat-Population (ITT); all randomized subjects who were dispensed medication and had at least one post-randomization visit
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Megestrol Acetate Oral Suspension Nanocrystal Dispersion | Megestrol Acetate Oral Suspension Micronized Formulation
Number analyzed (Participants) | 32 | 31
kg
  Overall | 5.4 (5.32) | 3.5 (4.03)
  Male | 7.0 (3.16) | 3.5 (4.72)
  Female | 2.3 (7.18) | 3.5 (3.42)

2. Secondary Outcome: Change From Baseline in Lean Mass
Time Frame: Baseline (Day 1) to Week 12
Population: Analysis is based on Intent-To-Treat-Population (ITT); all randomized subjects who were dispensed medication and had at least one post-randomization visit. Only 31 subjects were analyzed for the megestrol acetate oral suspension nanocrystal dispersion group based on available baseline measurements.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Megestrol Acetate Oral Suspension Nanocrystal Dispersion | Megestrol Acetate Oral Suspension Micronized Formulation
Number analyzed (Participants) | 31 | 31
kg | 2.1 (3.74) | 1.3 (2.82)

3. Secondary Outcome: Change From Baseline in Impedance
Description: Electrical impedance is a method for body composition assessment. The procedure involves sending a small current through the body and measuring the resistance in ohm. High resistance is associated with smaller amounts of fat-free mass. Smaller resistance is associated with large amounts of fat-free mass.
Time Frame: Baseline (Day 1) to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ohms
Arm/Group | Megestrol Acetate Oral Suspension Nanocrystal Dispersion | Megestrol Acetate Oral Suspension Micronized Formulation
Number analyzed (Participants) | 31 | 31
ohms | 21.6 (77.2) | 12.2 (54.2)

4. Secondary Outcome: Change From Baseline in Body Fat Mass
Time Frame: Baseline (Day 1) to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Megestrol Acetate Oral Suspension Nanocrystal Dispersion | Megestrol Acetate Oral Suspension Micronized Formulation
Number analyzed (Participants) | 31 | 31
kg | 3.2 (4.1) | 2.2 (3.4)

5. Secondary Outcome: Change in Hip Circumference
Time Frame: Baseline (Day 1) to Week 12
Population: Analysis is based on Intent-To-Treat-Population (ITT); all randomized subjects who were dispensed medication and had at least one post-randomization visit. Only 31 subjects and 29 subjects were analyzed, respectively based on available baseline measurements.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Megestrol Acetate Oral Suspension Nanocrystal Dispersion | Megestrol Acetate Oral Suspension Micronized Formulation
Number analyzed (Participants) | 31 | 29
cm | 2.5 (3.7) | 1.8 (3.6)

6. Secondary Outcome: Change in Waist Circumference
Time Frame: Baseline (Day 1) to Week 12
Population: Analysis is based on Intent-To-Treat-Population (ITT); all randomized subjects who were dispensed medication and had at least one post-randomization visit. Only 31 subjects were analyzed for the megestrol acetate oral suspension nanocrystal dispersion group based on available data measurements.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Megestrol Acetate Oral Suspension Nanocrystal Dispersion | Megestrol Acetate Oral Suspension Micronized Formulation
Number analyzed (Participants) | 32 | 31
cm | 7.1 (4.9) | 5.4 (4.7)

7. Secondary Outcome: Change in Tricep Skinfold
Time Frame: Baseline (Day 1) to Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Megestrol Acetate Oral Suspension Nanocrystal Dispersion | Megestrol Acetate Oral Suspension Micronized Formulation
Number analyzed (Participants) | 32 | 31
cm | 1.0 (2.6) | 1.5 (5.4)

8. Secondary Outcome: Change in Mid-arm Circumference
Time Frame: Baseline (Day 1) to Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Megestrol Acetate Oral Suspension Nanocrystal Dispersion | Megestrol Acetate Oral Suspension Micronized Formulation
Number analyzed (Participants) | 32 | 31
cm | -0.6 (11.5) | 1.1 (1.5)

9. Secondary Outcome: Change in Total Energy
Description: Food intake was quantified by the 24-hour recall food diary
Time Frame: Baseline (Day 1) to Week 12
Population: Analysis is based on Intent-To-Treat-Population (ITT); all randomized subjects who were dispensed medication and had at least one post-randomization visit. Only 27 subjects and 22 subjects were analyzed, respectively based on available baseline data.
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | Megestrol Acetate Oral Suspension Nanocrystal Dispersion | Megestrol Acetate Oral Suspension Micronized Formulation
Number analyzed (Participants) | 27 | 22
kcal | 215.9 (830.3) | 150.6 (1044.1)

10. Secondary Outcome: Quality of Life (QoL) Via Bristol-Myers Anorexia/Cachexia Recovery Instrument (BACRI) at Baseline (Day 3) and Week 12 (BACRI)
Description: The BACRI instrument is used to measure the benefit of weight gain treatment provided to anorexic patients on health related quality of life aspects. The scale is composed of 9 subscales (0 to 10 [worse to better]). The response was captured on a VAS scale in cm. The total BACRI score is the sum with a minimum score 0=worse and maximum score 90=better. These subscales are: change in weight impacting health; concern about weight; appearance change; change feeling of appearance; change in appetite; enjoy eating; overall feeling; benefit of treatment; and quality of life.
Time Frame: Baseline (Day 3) to Week 12
Population: Analysis is based on Intent-To-Treat-Population (ITT); all randomized subjects who were dispensed medication and had at least one post-randomization visit. Only 29 subjects were analyzed in the micronized formulation treatment group based on available baseline measurements.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Megestrol Acetate Oral Suspension Nanocrystal Dispersion | Megestrol Acetate Oral Suspension Micronized Formulation
Number analyzed (Participants) | 32 | 29
cm
  Baseline (Day 3) | 52.3 (9.38) | 50.1 (7.31)
  Week 12 | 67.6 (9.53) | 65.6 (14.78)

11. Secondary Outcome: Appetite at Baseline (Day 3) and Week 12
Description: Appetite was assessed via visual analogue scale (VAS) as part of the Bristol-Myers Anorexia/Cachexia Recovery Instrument (BACRI) (Question 5 only). The question was "To what extent has your appetite changed since the start of treatment?" The response was captured on a VAS scale in cm with a range from 0 ( "much worse") to 10 ("much better").
Time Frame: Baseline (Day 3) to Week 12
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Megestrol Acetate Oral Suspension Nanocrystal Dispersion | Megestrol Acetate Oral Suspension Micronized Formulation
Number analyzed (Participants) | 32 | 29
cm
  Baseline Day 3 | 6.1 (1.81) | 5.8 (1.16)
  Week 12 | 8.4 (1.30) | 8.0 (2.14)

ADVERSE EVENTS:
Time Frame: Approximately 16 weeks (baseline [day 1] through week 12 plus 30-day follow-up)
Groups:
- Megestrol Acetate Oral Suspension NanoCrystal Dispersion: Subjects were treated with 575 mg per day as single dose for 12 weeks
- Megestrol Acetate Oral Suspension Micronized Formulation: Subjects were treated with 800 mg per day as single dose for 12 weeks
Arm/Group | Megestrol Acetate Oral Suspension NanoCrystal Dispersion | Megestrol Acetate Oral Suspension Micronized Formulation
Serious Adverse Events (participants affected / at risk) | 14/32 | 14/31
Other Adverse Events (participants affected / at risk) | 30/32 | 30/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Megestrol Acetate Oral Suspension NanoCrystal Dispersion (N=32) | Megestrol Acetate Oral Suspension Micronized Formulation (N=31)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 2 (2)
Adrenal insufficiency (Endocrine disorders) | 3 (3) | 4 (4)
Adrenal suppression (Endocrine disorders) | 2 (2) | 2 (2)
Asthenia (General disorders) | 0 (0) | 1 (1)
Death of unknown cause (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Adrenal gland tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
HIV infection (Infections and infestations) | 0 (0) | 1 (1)
Meningitis tuberculous (Infections and infestations) | 0 (0) | 1 (1)
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 2 (2)
Blood cortisol abnormal (Investigations) | 6 (6) | 3 (3)
Blood cortisol decreased (Investigations) | 2 (2) | 0 (0)
Venous pressure jugular increased (Investigations) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Demyelinating polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Amenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Megestrol Acetate Oral Suspension NanoCrystal Dispersion (N=32) | Megestrol Acetate Oral Suspension Micronized Formulation (N=31)
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 2
Cardiac failure congestive (Cardiac disorders) | 3 | 2
Adrenal insufficiency (Endocrine disorders) | 4 | 8
Adrenal suppression (Endocrine disorders) | 4 | 2
Cushingoid (Endocrine disorders) | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Constipation (Gastrointestinal disorders) | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 4
Dyspepsia (Gastrointestinal disorders) | 6 | 2
Flatulence (Gastrointestinal disorders) | 3 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 3
Vomiting (Gastrointestinal disorders) | 0 | 4
Asthenia (General disorders) | 5 | 0
Non-cardiac chest pain (General disorders) | 1 | 3
Oedema peripheral (General disorders) | 1 | 3
Pyrexia (General disorders) | 2 | 4
Bronchitis (Infections and infestations) | 2 | 1
Gastroenteritis (Infections and infestations) | 2 | 3
Nasopharyngitis (Infections and infestations) | 2 | 1
Pharyngitis (Infections and infestations) | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 4
Urinary tract infection (Infections and infestations) | 3 | 1
Excoriation (Injury, poisoning and procedural complications) | 2 | 0
Alanine aminotransferase increased (Investigations) | 2 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 2
Blood cholesterol increased (Investigations) | 3 | 1
Blood cortisol abnormal (Investigations) | 4 | 2
Blood cortisol decreased (Investigations) | 3 | 4
Blood glucose increased (Investigations) | 1 | 2
Blood lactate dehydrogenase increased (Investigations) | 12 | 5
Blood triglycerides increased (Investigations) | 2 | 1
Cardiac murmur (Investigations) | 3 | 1
Low density lipoprotein increased (Investigations) | 3 | 0
Mean cell haemoglobin increased (Investigations) | 5 | 5
Mean cell volume increased (Investigations) | 8 | 5
Red blood cell count decreased (Investigations) | 5 | 2
Red cell distribution width increased (Investigations) | 9 | 5
Venous pressure jugular increased (Investigations) | 2 | 4
Anorexia (Metabolism and nutrition disorders) | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3
Dizziness (Nervous system disorders) | 1 | 2
Headache (Nervous system disorders) | 8 | 6
Paraesthesia (Nervous system disorders) | 0 | 2
Somnolence (Nervous system disorders) | 1 | 2
Tremor (Nervous system disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 3 | 1
Libido decreased (Psychiatric disorders) | 2 | 1
Amenorrhoea (Reproductive system and breast disorders) | 2 | 2
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Periorbital oedema (Skin and subcutaneous tissue disorders) | 2 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 3 | 2
Flushing (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 5 | 5
Systolic hypertension (Vascular disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All manuscripts, abstracts or other modes of presentation arising from the results of this study must be reviewed and approved in writing by Par, in advance of submission.